CLINICAL TRIAL: NCT02723903
Title: Efficacy of Hierarchical Treatment For Suspected Coronary Heart Disease Based on Somatization Symptom Checklist and Coronary Angiography
Brief Title: Hierarchical Treatment Based on Somatization Symptom Checklist
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81470391
Record Dates: First submitted 2016-02-15; First posted 2016-03-31 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Syndrome X
Keywords: somatization symptom score; SSS checklist; coronary angiography; Patient Health Questionnaire; Generalized Anxiety Disorder 7-items
MeSH Terms: conditions — Microvascular Angina | interventions — flupentixol, melitracen drug combination; Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- with CAD and somatic symptom (Other): Patients with the coronary artery disease and with the somatization symptom, the investigators treat the patients according to the guideline for coronary artery disease and anti-somatic agents (Deanxit, Prozac according to the somatization type)
  Interventions: Drug: Deanxit; Drug: Prozac; Procedure: coronary artery disease treatment
- without CAD, with somatic symptom (Other): Only somatic symptom is presented, anti-somatic agents is prescribed (Deanxit, Prozac according to the somatization type)
  Interventions: Drug: Deanxit; Drug: Prozac
- without CAD, without somatic symptom (No Intervention): Have neither coronary artery disease nor somatic symptom, continue follow-up.
- with CAD, without somatic symptom (Other): Patient with the coronary artery disease, without the somatization symptom, the investigators treat the patients according to coronary artery disease treatment guideline including coronary artery stent implantation,medication according to the severity of stenosis of the coronary arteries.
  Interventions: Procedure: coronary artery disease treatment

INTERVENTIONS:
Drug: Deanxit — we use Deanxit for the patient with anxiety
  Other Names: Deanxit as anti-anxiety treatment
  Arms: with CAD and somatic symptom; without CAD, with somatic symptom
Drug: Prozac — we use Prozac for the patient with depression
  Other Names: Prozac as anti-depression treatment
  Arms: with CAD and somatic symptom; without CAD, with somatic symptom
Procedure: coronary artery disease treatment — including medication, coronary artery stent implantation according to the severity of stenosis of the coronary arteries
  Other Names: re-vascularization
  Arms: with CAD and somatic symptom; with CAD, without somatic symptom

SUMMARY:
A comparative study is conducted on the patients with suspected coronary artery disease (CAD). The patient will undergo coronary angiography after a somatic symptom scale (SSS) survey is carried out combining with Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder 7-items (GAD-7). Patient is then treated according to the checklist score and coronary angiography result. The efficacy, sensitivity and specificity of the SSS checklist will be evaluated during following up.

DETAILED DESCRIPTION:
The presentation of physical complaints such as chest discomfort suggestive of suspicious coronary artery disease (CAD) but remain unexplained after negative finding from coronary angiography represents one of the most frustrating and puzzling problems in clinical medicine.A comparative study is conducted on the patients with suspected coronary artery disease. A somatic symptom scale (SSS) survey is carried out combining with Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder 7-items (GAD-7). Patient is treated according to the checklist score and coronary angiography result. Three surveys will be re-conducted 2 weeks after treatment. The sensitivity and specificity of the SSS checklist will be evaluated during following up.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected coronary artery disease

Exclusion Criteria:

* patients who have lost their self assessments of capacity.
* patients who have been previously confirmed serious mental disorders.
* patients who is taking anti-anxiety agents or anti-depression agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of somatization symptom score | 2 weeks after the first visit
  observe the efficacy by the score of somatic symptom scale (SSS), Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder 7-items (GAD-7)

SECONDARY OUTCOMES:
scale chest discomfort | 2 weeks after the first visit
  observe if the chest discomfort no change, alleviate or disappear
The efficacy of Patient Health Questionnaire | 2 weeks after the first visit
  observe the efficacy by the score of Patient Health Questionnaire (PHQ-9)
The efficacy of Generalized Anxiety Disorder 7-items | 2 weeks after the first visit
  observe the efficacy by the score of Generalized Anxiety Disorder 7-items (GAD-7)

CONTACTS AND LOCATIONS:
Overall Officials: Mao Jialiang, Docter, Study Chair — Renji hosipital,Jiaotong University, School of Medicine
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No